CLINICAL TRIAL: NCT04468178
Title: Clinical Results and RSA Migration Analysis of the GLOBAL ICON - Stemless Anatomic Shoulder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-RSA-Global-Icon-2020
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: osteoarthritis; shoulder; joint replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: prospective, randomized controlled mono-centric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shoulder prosthesis system GLOBAL ICON from DePuy (Experimental): The GLOBAL ICON stemless is a shaftless shoulder prosthesis system for anatomical reconstruction of the shoulder joint in cases of total or hemiarthroplasty in the shoulder. The base plate consists of titanium coated with hydroxyapatite, the head of cobalt-chrome.
  Interventions: Device: Total joint arthroplasty of the glenohumeral joint
- SIMPLICITY shoulder prosthesis system from Wright Medical (Active Comparator): The SIMPLICITY is a shaftless shoulder prosthesis system for anatomical reconstruction of the shoulder joint in cases of total or hemiarthroplasty in the shoulder. The base plate consists of titanium coated with hydroxyapatite, the head of cobalt-chrome.
  Interventions: Device: Total joint arthroplasty of the glenohumeral joint

INTERVENTIONS:
Device: Total joint arthroplasty of the glenohumeral joint — The arthroplasty of the glenohumeral joint will be performed as an anatomical reconstruction after primary or post-traumatic osteoarthritis.

SUMMARY:
The primary goal of the clinical trial is to determine that the GLOBAL ICON implant system from DePuy does not exhibit worse shoulder function after 2 years than the SIMPLICITY from Wright Medical. The primary endpoint is the Constant-Murley Shoulder Score (CMSS) of the implant after 2 years, the non-inferiority of which is to be demonstrated in comparison with an already established prosthetic system (SIMPLICITY, Wright Medical).

DETAILED DESCRIPTION:
The primary goal of the clinical trial is to determine that the GLOBAL ICON implant system from DePuy does not exhibit worse shoulder function after 2 years than the SIMPLICITY from Wright Medical. The primary endpoint is the Constant-Murley Shoulder Score (CMSS) of the implant after 2 years, the non-inferiority of which is to be demonstrated in comparison with an already established prosthetic system (SIMPLICITY, Wright Medical).

As secondary endpoints, the migration behavior of the humeral components over time will be determined by radiostereometric analysis (RSA), the further clinical-functional results and the satisfaction of the patients treated will be investigated. Clinical outcomes are measured using standardized and reproducible clinical scores (Oxford Shoulder Score -OSS and Short Form Health 36-SF-36 v1.0 ) at each time of examination.

Other endpoints include revision rate within the follow-up period, surgical time (incision to suture), and delays in surgical procedures due to instrumentation.

The times of data acquisition are the admission day before the operation to determine the preoperative status, the discharge day and the follow-up appointments after 3 months, 6 months, 12 months and 24 months to determine the postoperative status and course.

ELIGIBILITY:
Inclusion Criteria:

1. Trial participants need primary total shoulder replacement due to primary osteoarthritis or post-traumatic osteoarthritis
2. Trial participants are willing to take part in the clinical trial and intend to be available for the planned follow-up examinations.
3. Male, female and various subjects with age on the day of surgery from 18 to 80 years inclusive.
4. Subjects agree not to participate in any other clinical trial for at least 2 years (+ 3 weeks) using the index procedure. This includes clinical trials of medication, invasive procedures and medical devices. Questionnaire-based studies or other studies that are non-invasive and do not involve drug use are allowed.
5. Exclusion of intraoperative circumstances that require the implantation of a prosthesis type other than that provided for in the clinical trial (depending on the surgeon).

Exclusion Criteria:

1. Previous operation on the rotator cuff of the affected shoulder
2. Dysfunctional rotator cuff
3. Infection of the affected shoulder joint or systemic infection
4. Pregnant or breastfeeding women and those who are planning to become pregnant for up to 2 years (+3 weeks) using the index procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley Score (CMS) | 3 months postoperative
  The CMS covers different aspects of shoulder pathology: pain, activities of daily living, range of motion and strength. The possible maximum total score is 100 points (best function). Pain and activities of daily living are answered by the patient; range of motion and strength are answered by the orthopaedic surgeon.
Constant-Murley Score (CMS) | 12 months postoperative
  The CMS covers different aspects of shoulder pathology: pain, activities of daily living, range of motion and strength. The possible maximum total score is 100 points (best function). Pain and activities of daily living are answered by the patient; range of motion and strength are answered by the orthopaedic surgeon.
Constant-Murley Score (CMS) | 24 months postoperative
  The CMS covers different aspects of shoulder pathology: pain, activities of daily living, range of motion and strength. The possible maximum total score is 100 points (best function). Pain and activities of daily living are answered by the patient; range of motion and strength are answered by the orthopaedic surgeon.

SECONDARY OUTCOMES:
Oxford Shoulder Score (OSS) | 3 months postoperative
  The Oxford Shoulder Score (OSS) is a 12-item patient-reported questionnaire specifically designed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. Scores from each question are added so the overall score ranges from 12 to 60 with 12 being the best out-come.
Oxford Shoulder Score (OSS) | 12 months postoperative
  The Oxford Shoulder Score (OSS) is a 12-item patient-reported questionnaire specifically designed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. Scores from each question are added so the overall score ranges from 12 to 60 with 12 being the best out-come.
Oxford Shoulder Score (OSS) | 24 months postoperative
  The Oxford Shoulder Score (OSS) is a 12-item patient-reported questionnaire specifically designed for assessing outcomes of shoulder surgery e.g. for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. Scores from each question are added so the overall score ranges from 12 to 60 with 12 being the best out-come.
Short Form Health 36 (SF-36) | 3 months postoperative
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health consisting of eight scaled scores. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Short Form Health 36 (SF-36) | 12 months postoperative
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health consisting of eight scaled scores. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Short Form Health 36 (SF-36) | 24 months postoperative
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health consisting of eight scaled scores. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Smith, PD Dr., Principal Investigator — Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift
Locations (1):
- Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No